CLINICAL TRIAL: NCT03113916
Title: Culturally Competent Behavioral Intervention for Diabetes Risk Reduction
Brief Title: De Por Vida: A Diabetes Risk Reduction Intervention for Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01DK099277-04 (NIH)
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Diabetes; Weight Loss; PreDiabetes; Obesity
Keywords: Culturally-tailored; Weight Loss; Diabetes; Women; Hispanic; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss; Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: Trial participants are randomly assigned to one of two conditions: 1) Enhanced usual care control, or 2) a culturally tailored behavioral intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral (Experimental): 26 weekly behavioral intervention sessions 6 monthly behavioral intervention sessions Sessions focused on diet, physical activity, behavior change
  Interventions: Behavioral: Behavioural Lifestyle Intervention
- Enhanced usual care (No Intervention): Printed materials

INTERVENTIONS:
Behavioral: Behavioural Lifestyle Intervention — A culturally tailored behavioral intervention.
  Arms: Behavioral

SUMMARY:
This pragmatic randomized clinical trial will assess the efficacy, cost, and sustainability of a culturally tailored weight-loss program targeting obese Hispanic women with pre-diabetes or T2D. The intervention will be integrated into patient care at a Federally Qualified Health Center serving over 30,000 low-income patients, and will be delivered by trained clinic staff, with minimal support from research staff. After the effectiveness clinical trial, two cohorts of clinic patients will receive the intervention in a sustainability test.

DETAILED DESCRIPTION:
Hispanic women have the highest estimated lifetime risk of developing diabetes of all ethnic/gender groups in the US, and their prevalence rates of overweight and obesity are among the highest in the US. Currently, nearly 90% of Hispanic women aged 40-59 are overweight or obese. If diagnosed with Type 2 diabetes (T2D) at age 40, Hispanic women are projected to lose 12.4 life-years, and 21.5 quality-adjusted life-years.

Several clinical trials have produced compelling evidence demonstrating the benefits of weight-loss interventions for both diabetic and pre-diabetic individuals, but most of the successful interventions tested in large clinical trials have been too costly for implementation in community settings, and they have not been assessed under real life conditions, targeting vulnerable populations.

This study builds on the investigators' success with a culturally-tailored weight-loss intervention designed for Hispanic women. Elements of cultural adaptation will include: women-only groups, skill-building tasks around food measurement, focus on traditional dietary habits and cultural norms regulating food preparation and consumption, interactive learning formats with a minimum of written materials, culturally congruent physical activity, and addressing acculturative concerns.

Follow-up data, including change in weight, waist circumference, and diabetes outcomes, will be collected at 6-, 12-, and 18-months post randomization. Additional analyses will include the cost of delivering the intervention and assessing the intervention's sustainability. The results of this study will inform the development of interventions to prevent diabetes onset or manage T2D in this population.

Description of Measures Used

Southwest Food Frequency Questionnaire (SWFFQ).

The Southwestern Food Frequency Questionnaire (SWFFQ) consists of 158 food items and was adapted from the Arizona Food Frequency Questionnaire. It provides a culturally appropriate means of collecting dietary information for the Southwestern U.S. Hispanic populations predominantly of Mexican descent. It is the only Spanish bicultural and bilingual questionnaire in widespread use in the country. Examples of food items that are included in the questionnaire are nopalitos (cactus leaves), corn and flour tortillas, refried beans, machaca, and chorizo. The SWFFQ has been tested for validity and reliability (Taren et al, 2000). The output provides 87 nutrients in addition to 25 derived variables such as percent of calories from fat. VALIDATION PAPER Taren D, Tobar M, Ritenbaugh C, Graver E, Whitacre R, Aickin M. Evaluation of the Southwest Food Frequency Questionnaire. Ecology of Food and Nutrition 38:515-547, 2000.

General Practice Physical Activity Questionnaire (GPPAQ)

The GPPAQ is a validated screening tool for use in primary care that is used to assess adult (16 - 74 years) physical activity levels. It provides a simple, 4-level Physical Activity Index (PAI) categorizing patients as: Active, Moderately Active, Moderately Inactive, and Inactive. SOURCE: https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/192453/GPPAQ_-_guidance.pdf

Client Satisfaction Questionnaire (CSQ-8).

The CSQ-8 is a well-validated, 8-item Likert-type questionnaire that has been widely used in studies of physical and mental health among Spanish-speaking and Hispanic individuals. SOURCE http://www.csqscales.com/csq-8.htm

Barriers to Healthy Eating Questionnaire (BHEQ)

The BHE is a 22-item questionnaire asking individuals to rate various feelings or situations related to following the calorie and fat-restricted diet, eg, feelings of deprivation or cost of the recommended eating plan. It has 3 subscales: Emotions (11 items), Daily Mechanics of Following a Healthy Eating Plan (8 items), and Social Support (3 items). VALIDATION PAPER Impact of Perceived Barriers to Healthy Eating on Diet and Weight in a 24-Month Behavioral Weight Loss Trial. Wang, Jing et al. Journal of Nutrition Education and Behavior , Volume 47 , Issue 5 , 432 - 436.e1

Subjective Numeracy Scale

The Subjective Numeracy Scale (SNS) is a self-report measure of perceived ability to perform various mathematical tasks and preferences for the use of numerical versus prose information. The SNS has been validated against objective numeracy measures and found to predict comprehension of risk communications and ability to complete utility elicitations.

The De Por Vida study asked questions 3 and 4 of the SNS ability subscale which asked respondents to assess their numerical ability in different contexts. The scale contains no mathematics questions and has no correct or incorrect answers. VALIDATION PAPER Fagerlin, A., Zikmund-Fisher, B.J., Ubel, P.A., Jankovic, A., Derry, H.A., & Smith, D.M. Measuring numeracy without a math test: Development of the Subjective Numeracy Scale (SNS). Medical Decision Making, 2007: 27: 672-680.

Screening Questions for Limited Health Literacy

We asked 3 screening questions to assess limited health literacy validated by Chew et al. VALIDATION PAPER Chew LD, Griffin JM, Partin MR, et al. Validation of Screening Questions for Limited Health Literacy in a Large VA Outpatient Population. Journal of General Internal Medicine. 2008;23(5):561-566. doi:10.1007/s11606-008-0520-5.

Language-Based Acculturation Scale

A simple scale for quantifying English use among Mexican Americans was constructed from four brief questions which proved to have excellent scaling characteristics by Guttman Scalogram Analysis in two independent data sets. Construct validity was established by significant associations of the scale with ethnicity, place of birth, generation within the United States, and type of neighborhood. Highly significant associations were found between scale scores and use of oral contraceptives, parity, "fatalism" regarding health, and attitudes toward folk healers. These associations remained significant (though weak) after controlling for education and family income. The language scale thus appears to be reliable and valid, to be capable of distinguishing meaningful subsets among the Mexican American population, and to be applicable to health care investigation. VALIDATION PAPER A Simple Language-based Acculturation Scale for Mexican Americans: Validation and Application to Health Care Research. Deyo, Richard A.; And Others. American Journal of Public Health, v75 n1 p51-55 Jan 1985

ELIGIBILITY:
Inclusion Criteria:

* All participants will be patients who receive their primary medical care at the Virginia Garcia Memorial Health Center (VGMHC)
* Self-identified as Spanish-speaking Latina or Hispanic
* Female
* Age 18 and older
* BMI greater than or equal to 27kg/m2
* Classified as diabetic or prediabetic in the electronic medical record by at least one of the following:

  * Fasting plasma glucose ≥ 100
  * 2-h post glucose level on the 75-g oral glucose tolerance test ≥ 140-199 mg/dL (7.8-11.0 mmol/L)
  * Hemoglobin HBA1c ≥ 5.7
  * Diagnosis of diabetes in patient's medical chart
  * Diagnosis of prediabetes in patient's medical chart
* Residing in the Portland metropolitan area, and having no plans to leave the area in the next 18 months.
* Willing and able to attend the 26-weekly group meetings and 6 monthly group meetings.
* Willing to accept random assignment to the active intervention or enhanced usual care control.
* Clearance by the patient's VGMHC primary care physician to participate in the intervention.

Exclusion Criteria:

* Treatment for cancer in the past two years (excluding non-melanoma skin cancers).
* Having conditions that require limitation of physical activity or that would be contraindicated for the DASH (Dietary Approaches to Stop Hypertension) diet patterns.
* Taking weight-loss medication currently or within the past 6 months.
* Current or recent (< 12 months) pregnancy, breastfeeding, or planning pregnancy in the next 18 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 195 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nangel Lindberg, PhD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindberg NM, Vega-Lopez S, LeBlanc ES, Leo MC, Stevens VJ, Gille S, Arias-Gastelum M, Meenan R. Lessons Learned From a Program to Reduce Diabetes Risk Among Low-Income Hispanic Women in a Community Health Clinic. Front Endocrinol (Lausanne). 2021 Jan 8;11:489882. doi: 10.3389/fendo.2020.489882. eCollection 2020. PMID 33488511

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Intervention: 26 weekly behavioral intervention sessions 6 monthly behavioral intervention sessions Sessions focused on diet, physical activity, behavior change
  Behavioural Lifestyle Intervention: A culturally tailored behavioral intervention.
- Enhanced Usual Care: Printed materials and usual medical care
Period: Overall Study
Arm/Group | Behavioral Intervention | Enhanced Usual Care
Started | 99 | 96
Completed | 88 | 84
Not Completed | 11 | 12
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Pregnancy | 1 | 3
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral | Enhanced Usual Care | Total
Number analyzed (Participants) | 99 | 96 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 43 (10) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 96 | 195
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 96 | 195
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 96 | 195

OUTCOME MEASURES:

1. Primary Outcome: Weight in Kilograms
Description: Comparison of body weight trajectories in kilograms between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 99 | 96
kilograms
  Baseline | 87.1 [83.8 to 90.5] | 86.3 [82.9 to 89.7]
  6 Months | 84.4 [81.2 to 87.7] | 85.9 [82.6 to 89.2]
  12 Months | 84.2 [81.0 to 87.5] | 85.8 [82.5 to 89.2]
  18 Months | 84.2 [80.9 to 87.4] | 85.8 [82.5 to 89.1]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .001, Mixed Models Analysis; Slope = 2.63, 95% CI 2-sided [1.05 to 4.20]

2. Primary Outcome: Waist Circumference in Centimeters
Description: Comparison of waist circumference trajectories in centimeters between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Groups:
- Behavioral: Intervention
- Enhanced Usual Care: Control
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 99 | 96
centimeters
  Baseline | 115.2 [112.6 to 117.9] | 115.6 [112.8 to 118.2]
  6 months | 113.5 [110.9 to 116.1] | 114.7 [112.1 to 117.4]
  12 months | 112.9 [110.2 to 115.6] | 114.5 [111.7 to 117.2]
  18 months | 112.6 [109.8 to 115.4] | 114.3 [111.5 to 117.1]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .23, Mixed Models Analysis; Slope = -0.49, 95% CI 2-sided [-1.29 to 0.31]

3. Secondary Outcome: Hemoglobin HbA1c % (Transformed Using the Inverse Cube, or 1/HbAlc%^3)
Description: Comparison of hemoglobin HbA1c trajectories between the intervention and usual-care control groups.
  Because of the severe kurtosis and skewness present in this outcome, a transformation (using the inverse cube, or 1/HbAlc%^3) was undertaken to better meet the assumptions of the analysis. Thus, the trajectory differences between arms were formally tested using the inverse cube of HbA1c, and back transforming the least square mean estimates from this model will not result in the least square means in the original metric. We performed a sensitivity analysis using the untransformed HbA1c, and that model exhibited poorer model fit. We can present the crude, observed means, or the least square means from the model using the untransformed HbA1c if it is of greater priority to have more direct interpretability of the HbA1c values than using the model that better meets the statistical assumptions.
Time Frame: Baseline, 6, 12 and 18 months from enrollment
Population: Analysis limited to data available at different time points (6, 12, 18). As participants were required to come in to the clinic to collect their data it was challenging to get follow up data.
Measure: Least Squares Mean (95% Confidence Interval); unit: inverse cube of HbA1c percentage
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 99 | 96
inverse cube of HbA1c percentage
  Baseline | .00448 [.00413 to .00483] | .00445 [.00410 to .00481]
  6 Months | .00445 [.00410 to .00480] | .00439 [.00404 to .00474]
  12 months | .00437 [.00402 to .00472] | .00423 [.00388 to .00458]
  18 months | .00424 [.00388 to .00461] | .00397 [.00360 to .00434]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .06, Mixed Models Analysis; Slope = .000000676, 95% CI 2-sided [-.00000002 to .00000137]

4. Secondary Outcome: Fasting Blood Glucose (Fbg; Transformed Using the Inverse Square, or 1/Fbg in mg/dl^2 )
Description: Comparison of fasting blood glucose trajectories between the intervention and usual-care control groups.
  Because of the severe kurtosis and skewness present in this outcome, a transformation (using the inverse square, or 1/fasting blood glucose in mg/dl^2) was undertaken to better meet the assumptions of the analysis. Thus, the trajectory differences between arms were formally tested using the inverse square of fasting blood glucose, and back transforming the least square mean estimates from this model will not result in the least square means in the original metric. We performed a sensitivity analysis using the untransformed fasting blood glucose, and that model exhibited poorer model fit. We can present the crude, observed means, or the least square means from the model using the untransformed fasting blood glucose if it is of greater priority to have more direct interpretability of the fasting blood glucose values than using the model that better meets the statistical assumptions.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: inverse square of fbg mg/dl
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 99 | 96
inverse square of fbg mg/dl
  Baseline | .0000699 [.0000645 to .0000753] | .0000668 [.0000614 to .0000723]
  6 months | .0000699 [.0000645 to .0000752] | .000067 [.0000615 to .0000724]
  12 months | .0000695 [.0000641 to .0000748] | .0000676 [.0000622 to .000073]
  18 months | .0000685 [.0000617 to .0000752] | .0000692 [.0000625 to .000076]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .29, Mixed Models Analysis; Slope = -5.64, 95% CI 2-sided [-16 to 4.73] — Values given need to be multiplied by 10 to the power of -10 (i.e., x 10^-10)

5. Secondary Outcome: Total Cholesterol
Description: Comparison of total cholesterol trajectories between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 99 | 95
mg/dl
  Baseline | 195.6 [188.0 to 203.2] | 191.9 [184.1 to 199.7]
  6 months | 199.5 [192.3 to 206.7] | 193.8 [186.5 to 201.1]
  12 months | 203.5 [195.8 to 211.2] | 195.6 [187.9 to 203.4]
  18 months | 207.4 [198.4 to 216.5] | 197.5 [188.5 to 206.5]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .27, Mixed Models Analysis; Slope = .351, 95% CI 2-sided [-.277 to .978]

6. Secondary Outcome: Number of Fruit Servings Per Day (Transformed Using the Natural Log)
Description: Comparison of number fruit servings per day trajectories between the intervention and usual-care control groups.
  Because of the severe kurtosis and skewness present in this outcome, a transformation (using the natural log) was undertaken to better meet the assumptions of the analysis. Thus, the trajectory differences between arms were formally tested using the log of the number of fruit servings per day, and back transforming the least square mean estimates from this model will not result in the least square means in the original metric. We performed a sensitivity analysis using the untransformed number of fruit servings per day, and that model exhibited poorer model fit. We can present the crude, observed means, or the least square means from the model using the untransformed number of fruit servings per day if it is of greater priority to have more direct interpretability of the # of fruit servings per day values than using the model that better meets the statistical assumptions.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log of fruit servings per day
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
natural log of fruit servings per day
  Baseline | .637 [.410 to .795] | .511 [.352 to .671]
  6 months | .522 [.395 to .649] | .483 [.355 to .612]
  12 months | .406 [.271 to .542] | .456 [.319 to .594]
  18 months | .291 [.113 to .469] | .423 [.250 to .608]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .10, Mixed Models Analysis; Slope = -.015, 95% CI 2-sided [-.032 to .003]

7. Secondary Outcome: Number of Kilocalories
Description: Comparison of the number of kilocalories trajectories between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: kilocalories
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
kilocalories
  Baseline | 1546 [1435 to 1658] | 1431 [1319 to 1544]
  6 months | 1381 [1289 to 1473] | 1333 [1240 to 1426]
  12 months | 1215 [1117 to 1313] | 1234 [1135 to 1333]
  18 months | 1049 [924 to 1175] | 1135 [1009 to 1261]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = -11.2, 95% CI 2-sided [-23.0 to 0.7]

8. Secondary Outcome: Sugar Intake in Grams
Description: Comparison of the sugar intake in grams trajectories between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
grams
  Baseline | 79.9 [72.5 to 87.3] | 72.6 [65.2 to 80.1]
  6 months | 70.2 [64.1 to 76.3] | 66.7 [60.5 to 72.9]
  12 months | 60.5 [54.1 to 67.0] | 60.8 [54.2 to 67.3]
  18 months | 50.8 [42.5 to 59.1] | 54.8 [46.4 to 63.2]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .12, Mixed Models Analysis; Slope = -.63, 95% CI 2-sided [-1.41 to 0.16]

9. Secondary Outcome: Dietary Fiber Intake in Grams (Transformed Using the Natural Log)
Description: Comparison of the dietary fiber intake in grams trajectories between the intervention and usual-care control groups.
  Because of the severe kurtosis and skewness present in this outcome, a transformation (using the natural log) was undertaken to better meet the assumptions of the analysis. Thus, the trajectory differences between arms were formally tested using the log of the dietary fiber intake in grams and back transforming the least square mean estimates from this model will not result in the least square means in the original metric. We performed a sensitivity analysis using the untransformed dietary fiber intake in grams, and that model exhibited poorer model fit. We can present the crude, observed means, or the least square means from the model using the untransformed dietary fiber intake in grams if it is of greater priority to have more direct interpretability of the dietary fiber intake in grams values than using the model that better meets the statistical assumptions.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log of fiber intake in grams
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
natural log of fiber intake in grams
  Baseline | 3.15 [3.06 to 3.24] | 3.01 [2.92 to 3.10]
  6 months | 2.87 [2.80 to 2.95] | 2.90 [2.83 to 2.98]
  12 months | 2.87 [2.79 to 2.94] | 2.90 [2.83 to 2.98]
  18 months | 2.87 [2.79 to 2.94] | 2.90 [2.83 to 2.98]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .008, Mixed Models Analysis; Slope = .174, 95% CI 2-sided [.050 to .302]

10. Secondary Outcome: Saturated Fat Intake as Percentage of Total Energy Intake
Description: Comparison of the saturated fat intake as percentage of total energy intake trajectories between the intervention and usual-care control groups.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of total energy
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
Percentage of total energy
  Baseline | 9.13 [8.72 to 9.55] | 9.40 [8.98 to 9.82]
  6 months | 8.80 [8.45 to 9.15] | 8.98 [8.63 to 9.33]
  12 months | 8.47 [8.09 to 8.85] | 8.56 [8.18 to 8.94]
  18 months | 8.14 [7.66 to 8.62] | 8.14 [7.65 to 8.62]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .50, Mixed Models Analysis; Slope = .015, 95% CI 2-sided [-.029 to .059]

11. Secondary Outcome: Number of Vegetable Servings Per Day (Transformed Using the Natural Log)
Description: Comparison of the dietary intake of the number of vegetable servings per day trajectories between the intervention and usual-care control groups.
  Because of the severe kurtosis and skewness present in this outcome, a transformation (using the natural log) was undertaken to better meet the assumptions of the analysis. Thus, the trajectory differences between arms were formally tested using the log of the number of vegetable servings per day, and back transforming the least square mean estimates from this model will not result in the least square means in the original metric. We performed a sensitivity analysis using the untransformed outcome, and that model exhibited poorer model fit. We can present the crude, observed means, or the least square means from the model using the untransformed number of vegetable servings per day if it is of greater priority to have more direct interpretability of the outcome values than using the model that better meets the statistical assumptions.
Time Frame: Baseline, 6, 12, and 18 months
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log of vegetable servings / day
Arm/Group | Behavioral | Enhanced Usual Care
Number analyzed (Participants) | 98 | 96
natural log of vegetable servings / day
  Baseline | 1.37 [1.25 to 1.50] | 1.27 [1.15 to 1.40]
  6 months | 1.30 [1.20 to 1.40] | 1.20 [1.10 to 1.30]
  12 months | 1.22 [1.12 to 1.33] | 1.13 [1.02 to 1.24]
  18 months | 1.15 [1.01 to 1.29] | 1.05 [0.91 to 1.20]
Statistical Analysis 1: Comparison: Behavioral vs Enhanced Usual Care; Test type: Superiority; p = .99, Mixed Models Analysis; Slope = -.00003, 95% CI 2-sided [-.013 to .013]

12. Other Pre Specified Outcome: Average Program Cost Per Participant
Description: Average cost per participant of the De Por Vida intervention and enhanced usual care
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Behavioral Intervention | Enhanced Usual Care
Number analyzed (Participants) | 99 | 96
Dollars | 360.68 (63.01) | 0 (0)

13. Other Pre Specified Outcome: Recruit Participants for Sustainability Phase
Description: Number of participants recruited
Time Frame: Post-intervention for 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Sustainability Phase Participants: Participants recruited into sustainability groups
Arm/Group | Sustainability Phase Participants
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 6, 12 and 18 month assessment follow up time points.
Description: When an event was reported by a participant, study staff collected information on a form that asked for details about the event, and about ER, hospital and urgent care visits since the last assessment. An endocrinologist, blinded to study arm, then assessed whether the event was likely or unlikely to be study related and were monitored/assessed without regard to a specific Adverse Event Term and categorized after assessment. All events were reviewed by an independent safety monitor.
Arm/Group | Behavioral | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/98
Serious Adverse Events (participants affected / at risk) | 5/102 | 2/98
Other Adverse Events (participants affected / at risk) | 64/102 | 49/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=102) | Enhanced Usual Care (N=98)
Cholecystectomy (Gastrointestinal disorders) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Neurological (Nervous system disorders) | 1 (1) | 0 (0) — Neurological
Gynecological (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=102) | Enhanced Usual Care (N=98)
Gastrointestinal (Gastrointestinal disorders) | 7 (7) | 9 (9)
Hypoglycemia (Expected) (Endocrine disorders) | 12 (12) | 11 (11)
Infection (Infections and infestations) | 9 (9) | 17 (17)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 24 (24) | 12 (12)
Neurological (Nervous system disorders) | 6 (6) | 3 (3)
Urological (Renal and urinary disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03113916/Prot_SAP_000.pdf